CLINICAL TRIAL: NCT05096247
Title: Post Market Study To Collect Efficacy Data For The Treatment Of Wrinkles With A Radiofrequency Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cynosure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7027-PM01-2021
Record Dates: First submitted 2021-10-15; First posted 2021-10-27 (Actual); Results first posted 2023-11-28 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Wrinkle; Benign Pigmented Lesions; Benign Vascular Lesions

STUDY DESIGN:
Intervention Model Description: One site will enroll patients to be treated with the the RF device, and the other site will enroll patients to be treated with the RF device and the Intense Pulsed Light (IPL) laser.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Treatment with RF Device (Experimental): Subjects in this arm of the study will be treated with the radiofrequency device, and will receive up to 4 treatments on the face.
  Interventions: Device: TempSure
- Treatment with IPL and RF Device (Experimental): Subjects treated in this arm of the study will receive 2 treatments with just the radiofrequency device and then 2 treatments with both the radiofrequency and the IPL laser.
  Interventions: Device: TempSure; Device: Icon

INTERVENTIONS:
Device: TempSure — This device is an RF device.
Device: Icon — This device works with IPL (Intense Pulsed Light) handpieces.
  Arms: Treatment with IPL and RF Device

SUMMARY:
The intended use of the RF (radiofrequency) device used in this study is to assess the efficacy of the handpiece for the treatment of facial wrinkles. If the other device (Intense Pulsed Light) laser in this study is used, the intended use will be for the treatment of benign pigmented and/or vascular lesions.

ELIGIBILITY:
Inclusion Criteria:

* A healthy male or female 18 years of age or older.
* Agrees to be treated with the TempSure device.
* Understands and accepts obligation not to receive any other procedures on the treatment area through the length of the study.
* Understands and accepts the obligation and is logistically able to be present for all visits.
* Is willing to comply with all requirements of the study and sign the informed consent document.

Exclusion Criteria:

* Is pregnant or of childbearing potential and not using medically effective birth control, or has been pregnant in the last 3 months, currently breast feeding or planning a pregnancy during the study.
* The subject has a cut, wound, or infected skin on the area to be treated.
* The subject is on local, oral, or systemic anesthetic agents.
* The subject has nerve insensitivity to heat in the treatment area.
* The subject has any condition or is in a situation which in the investigators opinion may put the subject at significant risk, may confound study results or may interfere significantly with the subject's participation.

Exclusion Criteria for Icon Treatments Only:

* The subject is using systemic steroids (e.g. prednisone, dexamethasone) prior to or during the course of treatment.
* The subject has a medical condition or is receiving treatment that significantly compromise healing response.
* The subject has a history of light-induced seizures.
* The subject has a history of skin photosensitivity disorders.
* The subject has a history of hypertrophic scars or keloid formation.
* The subject has a history of radiation therapy in area to be treated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-09-03 (Actual); Primary Completion 2022-09-13 (Actual); Study Completion 2022-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Civiok, Study Director — Cynosure, Inc.
Locations (3):
- United States (3):
  - Cynosure, Westford, Massachusetts
  - Excellent Vision, Portsmouth, New Hampshire
  - Saluja Cosmetic and Laser Center, Huntersville, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gupta V, Sharma VK. Skin typing: Fitzpatrick grading and others. Clin Dermatol. 2019 Sep-Oct;37(5):430-436. doi: 10.1016/j.clindermatol.2019.07.010. Epub 2019 Jul 17. PMID 31896400

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment With RF Device | Treatment With IPL and RF Device
Started | 13 | 35
Completed | 13 | 35
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment With RF Device | Treatment With IPL and RF Device | Total
Number analyzed (Participants) | 13 | 35 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 33 | 45
  >=65 years | 1 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 32 | 44
  Male | 1 | 3 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 12 | 35 | 47
  Hispanic | 1 | 0 | 1
FitzPatrick Skin Type [Count of Participants; unit: Participants] — Fitzpatrick Skin Type is measured on a scale from I-VI, with I representing low amounts of melanin and VI representing high amounts of melanin. Additional details can be found in the article referenced in the reference section.
  Participants
    Fitzpatrick Skin Type I | 0 | 3 | 3
    Fitzpatrick Skin Type II | 6 | 11 | 17
    Fitzpatrick Skin Type III | 5 | 20 | 25
    Fitzpatrick Skin Type IV | 2 | 1 | 3
    Fitzpatrick Skin Type V | 0 | 0 | 0
    Fitzpatrick Skin Type VI | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Who Noticed Improvement
Description: Subjects graded themselves on a scale ranging from "Worsened" to "Very Much Improved" at the follow up visit. The number of subjects who graded themselves as "Improved" was reported.
Time Frame: 12 week follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment With RF Device | Treatment With IPL and RF Device
Number analyzed (Participants) | 13 | 35
Participants | 10 | 34

ADVERSE EVENTS:
Time Frame: Subjects had their adverse events collected throughout their participation in the study, approximately 12 months.
Description: Subjects treated in the RF + IPL device group did not have these adverse events broken down by device.
Arm/Group | Treatment With RF Device | Treatment With IPL and RF Device
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/35
Other Adverse Events (participants affected / at risk) | 13/13 | 5/35
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment With RF Device (N=13) | Treatment With IPL and RF Device (N=35)
Erythema (Skin and subcutaneous tissue disorders) | 13 | 5
Edema (Skin and subcutaneous tissue disorders) | 0 | 5
Bruising (Skin and subcutaneous tissue disorders) | 0 | 1
Crusting (Skin and subcutaneous tissue disorders) | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI cannot disclose confidential or proprietary information until after it becomes generally known or available to the public.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-20): https://cdn.clinicaltrials.gov/large-docs/47/NCT05096247/Prot_SAP_000.pdf